CLINICAL TRIAL: NCT04517552
Title: Investigation of Inflammation Using [C-11]-CS1P1
Acronym: CS1P1
Status: Active, not recruiting | Type: Observational
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology, Neuroradiology Section, Professor of Neurological Surgery, Director, Knight Alzheimer Research Imaging Program, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: IRB #202001057
Record Dates: First submitted 2020-07-08; First posted 2020-08-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental: [11C] CS1P1
  Interventions: Drug: [11C]-CS1P1

INTERVENTIONS:
Drug: [11C]-CS1P1 — Participants will receive a single intravenous bolus injection of 6.0 - 20.0 mCi (222-740 MBq) of the investigational radiotracer [11C] CS1P1. Participants will then undergo a [11C] CS1P1 PET/CT scan.

SUMMARY:
There is a compelling need for a noninvasive imaging approach to measure S1P1 in both preclinical models of diseases and humans. PET measures of S1P1 expression is critical for elucidating the pathophysiological roles of S1P1 in neuroinflammation and neurodegeneration. The relevance of S1P1 in clinical disease has become readily apparent with the FDA approval of the S1P1 modulator FTY720 (fingolimod) for treating relapsing-remitting MS (RR-MS). MS is a chronic autoimmune, inflammatory disease caused by lymphocytic infiltration that leads to demyelinating neurodegenerative disease.

DETAILED DESCRIPTION:
The primary objective of the initial IND study is to determine the safety of the [11C]-CS1P1 for PET imaging of S1P1 expression. The investigators will first complete whole-body PET dosimetry studies in healthy adult normal volunteers to calculate the actual radiation dose of each human organ and determine the allowable dose for a human subject when receiving a single dose for a PET scan. Second, complete imaging of the brain and lymph nodes of the neck in a wide range of ages of healthy adult normal control participants, both male and females to characterize [11C]-CS1P1 uptake in the brain and radiolabeled metabolite will be completed. Finally, a comparison of the normal control participants to patients with multiple sclerosis (MS) will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, any race;
2. Age ≥ 18 years;
3. Capable of providing written informed consent for volunteering to undergo research procedures.
4. Healthy volunteer or volunteer with a diagnosis of MS

Exclusion Criteria:

1. Hypersensitivity to [11C]-CS1P1 or any of its excipients;
2. Contraindications to PET, CT or MRI (e.g. certain incompatible electronic medical devices, inability to lie still for extended periods) that make it potentially unsafe for the individual to participate;
3. Severe claustrophobia
4. Women who are currently pregnant or breast-feeding;
5. Currently undergoing radiation therapy;
6. Any condition that, in the opinion of the Sponsor-Investigator or designee could increase risk to the participant, limit the participant's ability to tolerate the research procedures or interfere with collection of the data (e.g., renal or liver failure, advanced cancer);
7. Participants who in the last 6 months experienced any of the following cardiovascular conditions or findings in the screening electrocardiogram (ECG): unstable cardiac arrhythmias, myocardial infarction, unstable angina, stroke, transient ischemic attack or decompensated heart failure requiring hospitalization or Class III/IV heart failure;
8. Must not have participated in any clinical trial involving a study drug or device within the 30-days prior to study enrollment;
9. Must not participate in another drug or device study prior to the end of this study participation;
10. Current or recent (within 12 months prior to screening) participation in research studies involving radioactive agents such that the total research-related radiation dose to the participant in any given year would exceed the limits set forth in the U.S. Code of Federal Regulations (CFR) Title 21 Section 361.1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aim 1: Dosimetry/ Safety Group Ten healthy adult volunteers (5 males and 5 females) will be recruited and undergo whole-body PET/CT imaging for assessing the safety, dosimetry and metabolism of [11C]-CS1P1.
  Aim 2: Feasibility Cohort Aim 2A will consist of 24 adult volunteers that will be recruited and scanned to characterize [11C] CS1P1 uptake on PET scans of the brain and cervical lymph nodes, to assess for radiolabeled metabolites. Up to 20 participants who have completed Aim 2A will continue with the collection of test-retest and safety data, Aim 2B. Ten healthy controls age and gender-matched to 10 participants with MS will be invited to return for repeat imaging for test-retest reliability not less than 7 days after and not more than 12 months after baseline imaging.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
The tracer [11C]-CS1P1 will be injected for the first time into humans, using a dose range of 12-17 mCi for evaluations of safety, biodistribution, and dosimetry. | 2 years
  Whole-body PET/CT images (skull vertex to proximal thighs) will be obtained in 10 healthy volunteers (5 males and 5 females) for up to a maximum of 4 hours immediately following intravenous (IV) injection of 12-17 mCi of [11C]-CS1P1 (dosage range calculated from rodent dosimetry data extrapolated to humans).
PET imaging studies of [11C]-CS1P1 in healthy normal control participants and human participants with multiple sclerosis. | 2 years
  We hypothesize that specific binding of [11C]-CS1P1 is elevated in participants with neuroinflammatory/neurodegenerative diseases of the CNS compared to healthy normal control participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No